CLINICAL TRIAL: NCT03801161
Title: Influence of Inflammation on Micronutrient Status Assessment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: Newcastle University, UK (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PR-18006
Record Dates: First submitted 2018-03-29; First posted 2019-01-11 (Actual); Last update posted 2019-08-26 (Actual); Status verified 2018-09

CONDITIONS: Healthy Infants
Keywords: vitamin A; vitamin A isotope; vitamin D; ferritin; transferrin receptor; folate; cobalamin; beta-carotene; Inflammation
MeSH Terms: conditions — Inflammation | interventions — Hepatitis B Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy infants (No Intervention)
- Infants with an inflammatory condition (Experimental): Investigators will also use pentavalent (PENTA) vaccine as a means to induce controlled inflammation (closely mimic to natural infection). PENTA is a combination of five different vaccine antigens (Hepatitis B (HBV)/ Haemophilus influenza type b (Hib) / Tetanus-Diphtheria-whole cell Pertussis (TDwP)).
  Interventions: Biological: Pentavalent vaccine. It is a combination of five different antigens (Hepatitis B (HBV)/ Haemophilus influenzae type b (HiB) / Tetanus-Diphtheria-whole cell Pertussis (TDwP)).

INTERVENTIONS:
Biological: Pentavalent vaccine. It is a combination of five different antigens (Hepatitis B (HBV)/ Haemophilus influenzae type b (HiB) / Tetanus-Diphtheria-whole cell Pertussis (TDwP)). — Pentavalent vaccine is being recommended to provide infants at 6wk, 10wk and 14wk of age. This vaccine also induces plasma CRP >5 mg/L in infants within 24 hours of immunization.
  Arms: Infants with an inflammatory condition

SUMMARY:
Inflammation can influence several biochemical measurements those commonly used to interpret micronutrient status in children. Our primary objective is to investigate the effects of inflammation on several biochemical measurements used to interpret micronutrient status in children. A total of 40 infants (9-18 mo of age) will participate in this study. Investigators will use PENTA vaccines as a means to induce controlled inflammation (closely mimic to natural infection). PENTA is a combination of five different vaccine antigens (Hepatitis B (HBV)/ Haemophilus influenza type b (Hib) / Tetanus-Diphtheria-whole cell Pertussis (TDwP)). The investigators will also use two different stable isotopic retinols for the assessment of total body vitamin A stores. Baseline blood samples (5 mL) will be obtained from all infants and then randomly selected 30 infants will receive PENTA vaccines, while the other 10 infants will receive no vaccines. 24 hours after vaccination a finger-prick blood sample will be obtained from the infants in the vaccinated group to measure CRP and on the same day, blood samples (5 mL) will be obtained from infants who develop inflammation (CRP> 5mg/L) in the vaccine group and also from infants in the control group. Thus estimated plasma micronutrients and vitamin A stores before and after inflammation will calculate the effects of inflammation on the interpretation of micronutrient deficiencies based on biochemical indicator assessment.

DETAILED DESCRIPTION:
Background:

Subclinical micronutrient deficiencies remain a hidden aspect of malnutrition for which comprehensive data are lacking. Defining subclinical micronutrient deficiencies requires considering the prevalence of inflammation and its implications for the interpretation of micronutrient deficiencies based on biochemical indicator assessment. This study will provide a comprehensive profile of micronutrient status and antimicrobial resistance in a cohort of young children living in the densely populated urban slum.

Hypothesis:

I. Inflammation can influence several biochemical measurements those commonly used to interpret micronutrient status in children II. Micronutrient assessments can be performed successfully using finger/heel prick blood samples with microsamplers, thus increasing the ease of blood collection and reducing costs for cold storage and transport to the analytical laboratory.

Specific Objectives:

Our primary objective is to investigate the effects of inflammation on several biochemical measurements used to interpret micronutrient status in children. Our secondary aim is to test the applicability of a blood spot device allowing the determination of micronutrient status in field settings. Our exploratory objective is to make a comparative analysis of gut antimicrobial resistance genes (AMR) and resistome profile in children.

Methods:

A total of 40 infants (9-18 mo of age) will participate in this study. In this study, investigators will use two different stable isotopic vitamin A e.g., 13C10-retinyl acetate and 13C4-retinyl acetate. 400 μg of these isotopes, dissolved in 0.5 mL of sunflower oil, will be provided directly into the infant's mouth by using a direct replacement pipette. Mothers will be asked to breastfeed their infant after oral dosing to enhance absorption of the labeled vitamin A. Specific activity of 13C10- and 13C4- retinyl acetate in the blood samples will be measured by liquid chromatography-tandem mass spectrometry (LC/MS/MS). On the day of blood collection, a 24-h dietary recall and weekly morbidity questionnaires will be used. Investigators will also use PENTA vaccines as a means to induce controlled inflammation (closely mimic to natural infection). PENTA is a combination of five different vaccine antigens (Hepatitis B (HBV)/ Haemophilus influenza type b (Hib) / Tetanus-Diphtheria-whole cell Pertussis (TDwP)). This vaccination is beneficial to the infants since the World Health Organization recommends a booster vaccination dose. At the end of the study, PENTA vaccines will also be provided to the study infants in the "no-vaccine" group.

On day 0, all infants (n=40) will receive an oral dose of 13C10-retinyl acetate, and blood samples (5 mL) will be taken on day 4. On day 7 all infants (n=40) will also receive another oral dose of 13C4-retinyl acetate. 3-day later randomly selected 30 infants will receive PENTA vaccines (day 10), while the other 10 infants will receive no vaccines. 24 hours after vaccination a finger-prick blood sample will be obtained from the infants in the vaccinated group to measure CRP (QuikRead go, Orion, Finland). On the same day (day 11), blood samples (5 mL) will be obtained from infants who develop inflammation (CRP> 5mg/L) in the vaccine group and also from infants in the control group (day 11). Thus plasma micronutrients and vitamin A stores estimates on day 4 and day 11 will evaluate the effects of inflammation on the plasma micronutrient status indicators and total body vitamin A store. Blood microsamplers will be tested alongside venous blood collection to assess the feasibility of finger/heel prick sampling. Fecal samples, local surface water, and wastewater samples will be collected to test the prevalence of AMR resitomes in children and their environment.

Outcome measures/variables:

1. The following plasma biomarkers will be estimated before inflammation and 24 hours after inflammation

   * Inflammation markers: C-reactive protein (CRP) (mg/L) and α1-acid glycoprotein (AGP) (g/L)
   * Vitamin A status indicators: retinol (nmol/L), total body vitamin A stores (nmol), Retinol binding protein (RBP) (mg/L) and beta-carotene (nmol/L)
   * Iron status indicators: ferritin (ug/L) and soluble transferrin receptor (mg/L)
   * Folate/B12 status indicators: folate (nmol/L), methylmalonic acid (umol/L) and cobalamin (pmol/L)
   * Trace element status indicators: selenium (ug/L), copper (ug/L) and thyroglobulin (ug/L).
2. The usefulness of a microsampler device to collect blood samples for future micronutrient assessments.
3. Assessment and contrast of AMR gene abundances and diversity to develop resistomes

ELIGIBILITY:
Inclusion criteria:

1. 9 - 18 months of age
2. Infants with normal body temperature and normal CRP (<5 mg/L)
3. Infants receive breast milk from the mother at least once per day
4. Mothers produce a breast milk containing 30-40 nmol vitamin A /g milk fat
5. Infants received a high-dose vitamin A capsules at the time of the most recent national distribution campaign (within the last 2-4 months)
6. Mother is 18 - 45 years of age
7. Mother and her infant plan to stay in the study area for the duration of the study

Exclusion criteria:

1. Mother or infant has chronic disease
2. Mother or infant has acute illness on the day of data collection
3. Infant is anemic (Hb <90 g/L)
4. Infant has weight for length <80% of the reference median
5. Infants do not develop inflammation (CRP ≥5 mg/L) after PENTA vaccination

Ages: 9 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 75 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Inflammation marker C-reactive protein (CRP) levels in infants before and 1-day after inflammation | 24 hours
  In infants (9-18 mo) plasma CRP levels (mg/L) will be estimated by ELISA before and 24 hours after inflammation. Paired t-test will be used to evaluate the difference.
Vitamin A status in infants before and 1-day after inflammation | 24 hours
  In infants (9-18 mo) plasma retinol levels (nmol/L) will be estimated by HPLC before and 24 hours after inflammation.Paired t-test will be used to evaluate the difference.
Total body stores (TBS) of vitamin A in infants before and 1-day after inflammation | 24 hours
  In infants (9-18 mo) TBS of vitamin A (nmol) will be estimated before and 24 hours after inflammation. TBS will be measured by calculating the specific activities of 13C10- and 13C4- retinyl acetate in the blood samples by using liquid chromatography-tandem mass spectrometry (LC/MS/MS) method. Paired t-test will be used to evaluate the difference.
Iron status in infants before and 1-day after inflammation | 24 hours
  In infants (9-18 mo) plasma ferritin levels (ug/L) will be estimated by ELISA before and 24 hours after inflammation. Paired t-test will be used to evaluate the difference.
Iron status in infants before and 1-day after inflammation | 24 hours
  In infants (9-18 mo) plasma soluble transferrin receptor (sTfR) concentration (mg/L) will be estimated by ELISA before and 24 hours after inflammation. Paired t-test will be used to evaluate the difference.

CONTACTS AND LOCATIONS:
Locations (2):
- Bangladesh (2):
  - Clinical Trail Unit (CTU), icddr,b., Dhaka
  - Shaikh M Ahmad, Dhaka

IPD SHARING:
Plan to Share IPD: Undecided